CLINICAL TRIAL: NCT03493100
Title: Influence of Oral Nutritional Supplementation in Geriatric Fracture Patients on Muscle Functionality, Quality of Life and Nutritional Status
Brief Title: Hohenheim Malnutrition Study in Geriatric Fracture Patients
Acronym: HohMal2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HohMal2
Record Dates: First submitted 2017-06-21; First posted 2018-04-10 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-04

CONDITIONS: Geriatric Patients
Keywords: oral nutritional supplementation; geriatrics; bone fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral nutritional supplementation (Experimental): This group receives optimized nutritional support, by ONS for a period of four weeks.
  Interventions: Dietary Supplement: oral nutritional supplementation
- Control (Other): The control group will receive treatment according to usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Dietary Supplement: oral nutritional supplementation — The intervention group will receive optimized nutritional support, by ONS. While hospitalized each patient receives 2 portions of oral supplementation per day. For remaining days supplementation is calculated individually according to a sarcopenia/energy balance schema resulting in none or maximum 2 portions per day.
  Arms: oral nutritional supplementation
Other: Usual care — The control group will receive treatment according to usual care.
  Arms: Control

SUMMARY:
The aim of this study is to evaluate long-term effects of early and prolonged individualized and optimized nutritional support using ONS for four weeks, in combination with a defined physiotherapy regimen, on sarcopenia and other outcome parameters in elderly fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 75 years, or
* age ≥ 65 years and Carlson-Comorbidity-Index of ≥ 5 and
* written informed consent

Exclusion Criteria:

* progressive cancer disease
* relevant pre-existing chronic conditions (in order to avoid disease related impact on outcome parameters)
* insufficient German speech intelligibility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
hand grip strength | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  The primary endpoint is the change in muscle functionality of the study groups after 4 weeks by the measurement of hand grip strength using Jamar®-Dynamometer.

SECONDARY OUTCOMES:
Nutritional status | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up. Measured using Mini Nutritional Assessment (MNA).
Mobility | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up. Measured using Elderly Mobility Scale (EMS).
Arm/leg circumference | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Extracellular to body cell mass ratio (ECM/BCM - Ratio) | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Skinfold thickness | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Quality of life | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up. Measured using Activity of daily living (ADL) questionnaire and EQ-5-DL questionnaire.
Comorbidity rate | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Medical condition | Participants will be followed from day 1 to day 180.Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks.
Sarcopenia prevalence | Participants will be followed from day 1 to day 180.Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks.
Phase angle | Participants will be followed from day 1 to day 180. Examinations take place at discharge, after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Routine laboratory tests (serum plasma) | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Vitamin D in serum | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference in blood serum between intervention and control group at discharge and after 4 weeks follow-up.
Vitamin B12 in serum | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference in blood serum between intervention and control group at discharge and after 4 weeks follow-up.
Folic acid in serum | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference in blood serum between intervention and control group at discharge and after 4 weeks follow-up.
CRP (C-reactive protein) in serum | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference in blood serum between intervention and control group at discharge and after 4 weeks follow-up.
BCM (body cell mass) | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
Body weight | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.
BMI (body mass index) | Participants will be followed from day 1 to day 180. Examinations take place after 4 weeks, after 3 months and after 6 months.
  Difference between intervention and control group at discharge and after 4 weeks follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Principal Investigator — University of Hohenheim
Locations (1):
- University of Hohenheim, Stuttgart, Germany